CLINICAL TRIAL: NCT00491023
Title: Examining Macrophage Influx and Vascularization in Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0075
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2007-02

CONDITIONS: Pancreatitis; Diabetes
MeSH Terms: conditions — Pancreatitis; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Our aim in this study is to find out if we can locate the similar reduction in the recruitment of macrophages, remodeling of vasculature and do they correlate in the number and area of the islets in pancreas as in the mouse model.

ELIGIBILITY:
Inclusion Criteria:

* Pancreas tissue sections from preparates from pancreatic surgery.
* Patients having chronic pancreatitis with or without diabetes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-02; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James DeGregori, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Aurora, Colorado, United States